CLINICAL TRIAL: NCT01078714
Title: Study of the Efficiency of a Treatment by Bumetanide in a Population of Autistic Children
Brief Title: Efficiency of Bumetanide in Autistic Children
Acronym: BUMEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RB09-017
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Autistics Children
Keywords: Autism; Bumetanide; GABA; NKCC1
MeSH Terms: conditions — Autistic Disorder | interventions — Bumetanide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bumetanide (Experimental)
  Interventions: Drug: bumetanide
- Control (Placebo Comparator)
  Interventions: Drug: bumetanide

INTERVENTIONS:
Drug: bumetanide — Administration by oral route in 2 times (in the morning and evening) of 0.5 mg by taking (= 1 mg by 24 hours)

SUMMARY:
The purpose of this study is to determine if a treatment by bumetanide presents an efficiency at the level of the neuronal maturation in the autism

ELIGIBILITY:
Inclusion Criteria:

* Children from 3 to 10 years old, answering the diagnosis of typical autism according to the diagnostic criteria of autism of the classification of the WHO ( CIM-10) and the parents of which gave a free, enlightened and written consent.

Exclusion Criteria:

* Patients epileptic autistics treated by anticomitiaux or having hurts of the central nervous system
* Patients autistics receiving a psychotropic treatment
* Patients presenting disorders electrolytes
* Patients presenting a hypersensibility known about sulpha drugs
* Presenting patients against indications relative to the treatment by bumetanide
* Patients already treated by diuretics
* Patients presenting a hepatic or renal incapacity
* Patients presenting an elongation of the QT to the electrocardiogram.
* Patients autistics of CARS sore is lower than 30.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Child Autism Rating Scale score | day 0 to day 90

SECONDARY OUTCOMES:
Clinical global impressions score | day 0 to day 90
Repetitive end restricted behavior score | day 0 to day 90
GRAM score | day 0 to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Eric LEMONNIER, Dr, Principal Investigator — CHRU de Brest
Locations (3):
- France (3):
  - Lemonnier, Brest
  - Chevreuil, Rennes
  - DUPIN, Vannes

REFERENCES:
- [Derived] Lemonnier E, Degrez C, Phelep M, Tyzio R, Josse F, Grandgeorge M, Hadjikhani N, Ben-Ari Y. A randomised controlled trial of bumetanide in the treatment of autism in children. Transl Psychiatry. 2012 Dec 11;2(12):e202. doi: 10.1038/tp.2012.124. PMID 23233021